CLINICAL TRIAL: NCT03352960
Title: Environment and Childhood Project Based on a Multicentric Mother-child Cohort of Spain
Acronym: INMA
Status: Active, not recruiting | Type: Observational
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Jesus Ibarluzea, Principal Investigator, Basque Health Service
Other Study IDs: 22090111
Record Dates: First submitted 2017-11-10; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Pollutant Effects in the Growth and Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
INMA - INfancia y Medio Ambiente [Environment and Childhood] Project is a research network of several Spanish groups that created a project with the aim to study the paper of the more relevant environmental pollutants in the air, water and diet during the pregnancy and beginning of life, and their effects in the growth and development.

The INMA Project is based on the experience acquired by groups that studied several cohorts with different objectives: the cohort of Riera d'Ebre (n=102), an area with high levels of organochlorine compounds and mercury, evaluated the relationship between these exposures and the neurological development of the children; the cohort of Menorca (n=492), studied the relationship between the early exposure to irritating of the air and allergens with the development of allergy and asthma; and the cohort of Granada (n=668), that studied the incidence of reproductive disorders in men in relation to the exposure to endocrine disruptors.

Based on the experience of these previous cohorts, other 4 new cohorts were designed to evaluate the impact of environmental exposures in children's health: Valencia (n=787), Sabadell (n=622), Asturias (n=485) and Gipuzkoa (n=612), that followed the same protocol. The population of the study are pregnant women of the general population who lived in each area of study (Ribera d' Ebre, Menorca, Granada, Valencia, Sabadell, Asturias, and Gipuzkoa and their children. Each cohort had different periods and types from recruitment. In the cohorts of Ribera d'Ebre and Granada, the mothers were recruited during the admission to the hospital at the moment of the childbirth. In Ribera d'Ebre, the recruitment was between March 1997 and December 1999, whereas in Granada it was between October 2000 and July 2002. In Menorca, all the eligible women who went to the prenatal visit in some of the sanitary centres of the island (private or public) were invited to participate in the study, and the recruitment lasted a year starting in July 1997. In the 4 new cohorts the recruitment took place during the first prenatal visit (between weeks 10 and 13 of gestation) in the public hospital of reference or in the health centre of the area. The periods of recruitment went from February 2004 to June 2005 in Valencia, from July 2004 to July 2006 and May 2007 to July 2007 (there was an additional round of recruitment) in Sabadell, from May 2004 to June 2007 in Asturias, and from April 2006 to January 2008 in Gipuzkoa.

ELIGIBILITY:
Inclusion Criteria:

To belong to the study area (specific of each cohort). To be minimum 16 years. To have a unique pregnancy To give birth in the reference hospital

Exclusion Criteria:

To have followed any program of assisted reproduction To have communication problems

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The mothers were recruited between 1999 and 2008. The recruitment took place during the first prenatal visit (between weeks 10 and 13 of gestation) in the public hospital of reference or in the health centre of the area. The pregnant women included in the study were: Ribera d'Ebre (n=102), Menorca (n=492), Granada (n=668), Valencia (n=787), Sabadell (n=622), Asturias (n=485) and Gipuzkoa (n=612).
Sampling Method: Non-Probability Sample
Enrollment: 2957 (Actual)
Dates: Start 1997-01 (Actual); Primary Completion 2010-09-28 (Actual); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Development | 4 years
  BMI (kg/m^2)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Public Health, San Sebastián, Gipuzkoa, Spain